CLINICAL TRIAL: NCT03590236
Title: Graded Exposure Therapy in Women With Chronic Pelvic Pain
Brief Title: Graded Exposure Therapy in Chronic Pelvic Pain
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Universidad de Granada (Other)
Responsible Party: Principal Investigator, Marie Carmen Valenza, Principal investigator, Universidad de Granada
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DF0069UG
Record Dates: First submitted 2017-09-07; First posted 2018-07-18 (Actual); Last update posted 2018-07-18 (Actual); Status verified 2018-07

CONDITIONS: Chronic Pelvic Pain
Keywords: women; chronic pelvic pain; fear avoidance
MeSH Terms: interventions — Implosive Therapy; Physical Therapy Modalities

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Graded exposure therapy (Experimental): Patients in this group received graded exposure therapy added to physiotherapy
  Interventions: Other: Graded exposure therapy
- Physiotherapy (Active Comparator): Patients included in this group received the standard treatment based on a physiotherapy approach.
  Interventions: Other: Physiotherapy
- Control group (No Intervention): Waiting list patients

INTERVENTIONS:
Other: Graded exposure therapy — Patients included in this group received graded exposure therapy consisting on counselling, a graded activity through postural exercises and individual training focused on 5 activities selected by the patients. The treatment will include 5 sessions added to the 12 sessions of physiotherapy.
  Other Names: Exposure therapy
  Arms: Graded exposure therapy
Other: Physiotherapy — Physiotherapy intervention will include soft tissue mobilizations and myofascial release combined with deep-pressure massage to decrease trigger point-related pain and tension. In addition joint mobilization and muscle energy techniques will be included.
  Arms: Physiotherapy

SUMMARY:
Chronic pelvic pain (CPP) is considered as nonmalignant recurrent or continuous pain related to the structures of the pelvis. The objective of this study was to evaluate the effects of graded exposure therapy in women with chronic pelvic pain.

DETAILED DESCRIPTION:
Chronic pelvic pain (CPP) is considered as nonmalignant recurrent or continuous pain related to the structures of the pelvis. This condition lasts at least 6 months, and many times is associated with negative cognitive, emotional, sexual and behavioral consequences.In addition to the high economic cost, CPP is also costly in emotional and psychological suffering. This clinical trial aims to evaluate the effects of a program based on graded exposure therapy in women with chronic pelvic pain.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of chronic pelvic pain
* Moderate fear of movement

Exclusion Criteria:

* Other clinical diagnosis.
* Men
* Other pathology such as neurological disease.
* Cognitive impairment.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2017-08-20 (Actual); Primary Completion 2018-02-12 (Actual); Study Completion 2018-08-10 (Estimated)

PRIMARY OUTCOMES:
Fear-avoidance behaviors | Baseline, 6 weeks
  Changes from baseline to the end of the intervention will be assessed with the Fear Avoidance Beliefs Questionnaire (FABQ) using the physical activity subscale. This subscale focus on patients' beliefs about how physical activity affected their pain. The values ranges from 0 to 24 with higher scores indicating higher levels of fear-avoidance beliefs.

SECONDARY OUTCOMES:
Pain assessed by the Brief Pain Inventory | Baseline, 6 weeks
  Changes from baseline to the end of the intervention on pain will be assessed using the Brief Pain Inventory. This instrument evaluates the intensity of pain and also the degree to which the pain interferes in activities of daily living. The arithmetic mean ranging from 0 to 10 of the four severity items will be used as measures of pain severity; the arithmetic mean ranging from 0 to 10 of the seven interference items will be used as a measure of pain interference. Higher score represents worse pain.
Disability | Baseline, 6 weeks
  Changes from baseline to the end of the intervention will ibe assessed using the Oswestry Disability Index. It includes 10 items that assess how pain affects common daily activities. Scores range from 0 (no disability) to 100 (completely disabled), so higher scores indicate higher disability.
Activity performance | Baseline, 6 weeks
  The perceived quality of performance will be assessed using the Canadian Ocuppational Performance Measure

CONTACTS AND LOCATIONS:
Overall Officials: Marie CArmen Valenza, PhD, Principal Investigator — Universidad de Granada
Locations (1):
- Department of Physical Therapy, Granada, Spain

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Ariza-Mateos MJ, Cabrera-Martos I, Ortiz-Rubio A, Torres-Sanchez I, Rodriguez-Torres J, Valenza MC. Effects of a Patient-Centered Graded Exposure Intervention Added to Manual Therapy for Women With Chronic Pelvic Pain: A Randomized Controlled Trial. Arch Phys Med Rehabil. 2019 Jan;100(1):9-16. doi: 10.1016/j.apmr.2018.08.188. Epub 2018 Oct 9. PMID 30312595